CLINICAL TRIAL: NCT04466696
Title: Feasibility of ERAS Protocol in T4 Colorectal Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, Head of Department, University of Rome Tor Vergata
Other Study IDs: 3
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: T4 Colorectal Cancer; ERAS; Colon Cancer; Fast Track Protocol
Keywords: colon cancer; ERAS; fast track; t4 colorectal cancer; colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- t4 colorectal cancer treated with ERAS protocol: prospective from January 2016 to May 2020
  Interventions: Behavioral: ERAS protocol
- t4 colorectal cancer treated with standards of care: retrospective from January 2010 to December 2015

INTERVENTIONS:
Behavioral: ERAS protocol — items of ERAS protocol applied
  Groups: t4 colorectal cancer treated with ERAS protocol

SUMMARY:
Patients diagnosed with T4 colorectal cancer represent a specific subgroup of colorectal patients, frequently composed of fragile patients whose advanced nature of the disease often requires a multi organ resection by an open surgery approach and frequently leads to higher intra/postoperative complication.Those characteristics makes them to be considered less suitable for ERAS protocol, especially regarding an expected difficult compliance to postoperative items.

The impact of enhanced recovery program on postoperative outcomes in this subset of patients has never been addressed in literature, in fact most of studies either excluded T4 patients due to higher rates of complication or adopted an homogeneous patient sampling analizing all stage colorectal cancer together.

Our aim is to investigate the feasibility of ERAS protocol in T4 colorectal patient, primary outcome was to compare postoperative lenght of stay between T4 colorectal patients treated with ERAS protcol and those treated with standard of care.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cacer
* hystologic diagnosis of adenocarcinoma of the colon/rectum
* clinically staged T4
* written informed consent to surgery obtained

Exclusion Criteria:

* pregnancy
* failure to perform colonic or rectal resection
* synchronous cancer at time of colorectal cancer diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical diagnosis of stage T4 colorectal cancer who underwent surgical resection between January 2016 to January 2020 at Minimally Invasive Surgery Unit of Tor Vergata University Hospital were prospectively enrolled in the ERAS group and treated with fast track protocol. Postoperative short outcomes were compared to a control group treated with conventional care that underwent surgical resection for T4 colorectal cancer at the same center from January 2010 to December 2015. Data of the control group were collected retrospectively from a prospectively mantained database.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay | 30 days
  number of days from surgery to discharge